CLINICAL TRIAL: NCT03702335
Title: Impact of Comprehensive Dietary Counseling on Dietary Quality, Mental Health, and Quality of Life in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Jung Eun Kim, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: S3
Record Dates: First submitted 2018-10-05; First posted 2018-10-11 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Aging; Age Problem; Age-related Cognitive Decline; Age-Related Atrophy
Keywords: Older adults; Dietary consultation; Mental health; Sleep quality; Dietary quality; Cardio-metabolic health
MeSH Terms: conditions — Psychological Well-Being; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Counselling (Experimental): Each subject will receive a comprehensive dietary counselling for the first 12-weeks of the study, which will be followed by another 12-weeks without dietary counselling.
  Interventions: Behavioral: Dietary Counselling
- No Dietary Counselling (No Intervention): Subjects in the control group will be followed for 24-weeks without any dietary counselling.

INTERVENTIONS:
Behavioral: Dietary Counselling — Intervention group will be given a comprehensive dietary guidance on how to choose healthier options when eating out, as well as how to personally prepare a healthy meals.
  Arms: Dietary Counselling

SUMMARY:
As a person ages, an incidence of mental distress such as depression and anxiety increases while the quality of life decreases. Singapore's population is aging rapidly and older adults may suffer from mental distress and deteriorated quality of life. Recent evidence suggests that good nutrition is essential for mental health and quality of life in older adults.

Previous research reported that provision of nutrition education and cooking workshops to people with mental illness for 3 months achieved healthy dietary change and improved mental health. This proposed study aims to further assess the effect of comprehensive dietary counselling on dietary quality, cardio-metabolic, mental health, sleep quality, and quality of life through a 24-wk parallel intervention study in Singapore older adults.

The investigators hypothesised that older adults who receive comprehensive dietary counselling will improve dietary quality, cardio-metabolic health, mental health, sleep quality, and quality of life when compared to older adults who do not receive comprehensive dietary counselling.

DETAILED DESCRIPTION:
Fifty female Chinese older adults (aged 60+y) will be recruited with the expectation that ≥ 40 subjects will complete the study. This is a 24-wk parallel, single-bind, prospective study design with subjects randomly assigned to either receiving comprehensive dietary counselling (intervention group) or not receiving comprehensive dietary counselling (control group). Subjects in the intervention group will only receive comprehensive dietary counselling for first 12-wk and then they will be followed for another 12-wk without comprehensive dietary counselling. Subjects in the control group will be followed for 24-wk without any intervention. Dietary quality, mental health, sleep quality, daily physical activity and quality of life will be assessed and blood lipid-lipoproteins, glucose and insulin concentrations will be measured from the collected blood samples.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give an informed consent
2. Age ≥60 years
3. No weight change >3kg in the past 3 months
4. Not exercising vigorously over the past 3 months
5. Does not have any intestinal disorders, including lactose intolerance
6. No acute illness
7. Non-smoker
8. Non-vegetarian
9. Not drinking more than 2 alcoholic drinks/day
10. Not taking any lipid-lowering and blood pressure controlling medications less than 3 years

Exclusion Criteria:

1. Unable to give an informed consent
2. Age < 60 years
3. Weight change >3kg in the past 3 months
4. Exercises vigorously over the past 3 months
5. Have intestinal disorders, including lactose intolerence
6. Having acute illness
7. Smoking
8. Vegetarian
9. Drinking more than 2 alcoholic drinks/day
10. Taking lipid-lowering and blood pressure controlling medications less than 3 years

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 50 (Estimated)
Dates: Start 2018-11-13 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Change in diet | Every 2 week for the first 12 weeks and every 4 weeks for the last 12 weeks (Week 0, week 2, week 4, week 6, week 8, week 10, week 12, week 16, week 20, week 24)
  Dietary assessment, 3-day food record (participant)
Change in mental health status | Every 4 weeks (Week 0, week 4, week 8, week 12, week 16, week 20 and week 24)
  Mental Health Questionnaire - Consisting of basic health screen recording anthropometric measurements, visual functioning questionnaire scale (1; Good, 2; Acceptable, 3; Poor), Lifestyle (0; Never, 1; 1-3 times/month, 2; 1-3 times/week, 3; 4-6 times/week, 4; daily), depression scale (Yes or no questionnaire)
Change in quality of life | Every 4 weeks (Week 0, week 4, week 8, week 12, week 16, week 20 and week 24)
  Quality of Life Questionnaire
  * Subjective scale rating (1; very dissatisfied, 2; dissatisfied, 3; neither satisfied not dissatisfied, 4; satisfied, 5; very satisfied) assessing quality of life, health and other areas of life.
Change in sleep quality | Every 4 weeks (Week 0, week 4, week 8, week 12, week 16, week 20 and week 24)
  Pittsburgh Sleep Quality Assessment (PSQI) - Recall based questionnaire assessing sleep habits for the past one month only which includes sleeping timing habits and quality of sleep (Very good, Fairly good, Fairly bad and very bad)

SECONDARY OUTCOMES:
Change in diet | Every 12 weeks (Week 0, week 12 and week 24)
  Dietary Assessment, 3-day food record (Participant's family member)
Change in weight | Every 4 weeks (Week 0, week 4, week 8, week 12, week 16, week 20 and week 24)
  Weight (kg)
Change in waist circumference | Every 4 weeks (Week 0, week 4, week 8, week 12, week 16, week 20 and week 24)
  Waist Circumference (cm)
Change in blood pressure | Every 4 weeks (Week 0, week 4, week 8, week 12, week 16, week 20 and week 24)
  Systolic and diastolic blood pressure (mmHg) after a 10 hour overnight fast
Change in total cholesterol | Every 12 weeks (Week 0, week 12, and week 24)
  Total cholesterol (mmol/l)
Change in high-density lipoprotein cholesterol | Every 12 weeks (Week 0, week 12, and week 24)
  High-density lipoprotein cholesterol (mmol/l)
Change in low-density lipoprotein cholesterol | Every 12 weeks (Week 0, week 12, and week 24)
  Low-density lipoprotein cholesterol (mmol/l)
Change in total triglyceride | Every 12 weeks (Week 0, week 12, and week 24)
  Total triglyceride (mmol/l)
Change in blood glucose concentration | Every 12 weeks (Week 0, week 12, and week 24)
  Blood glucose concentration
Change in blood insulin concentration | Every 12 weeks (Week 0, week 12, and week 24)
  Blood insulin concentration
Change in daily physical activity | Daily (Week 0 to week 24)
  Tracked with an electronic activity tracker

CONTACTS AND LOCATIONS:
Overall Officials: Jung Eun Kim, PhD, RD, Principal Investigator — National University of Singapore
Locations (2):
- Singapore (2):
  - National University of Singapaore, Singapore
  - Hannah Senior Activity Centre, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Parletta N, Zarnowiecki D, Cho J, Wilson A, Bogomolova S, Villani A, Itsiopoulos C, Niyonsenga T, Blunden S, Meyer B, Segal L, Baune BT, O'Dea K. A Mediterranean-style dietary intervention supplemented with fish oil improves diet quality and mental health in people with depression: A randomized controlled trial (HELFIMED). Nutr Neurosci. 2019 Jul;22(7):474-487. doi: 10.1080/1028415X.2017.1411320. Epub 2017 Dec 7. PMID 29215971
- [Result] Bogomolova S, Zarnowiecki D, Wilson A, Fielder A, Procter N, Itsiopoulos C, O'Dea K, Strachan J, Ballestrin M, Champion A, Parletta N. Dietary intervention for people with mental illness in South Australia. Health Promot Int. 2018 Feb 1;33(1):71-83. doi: 10.1093/heapro/daw055. PMID 27476869
- [Derived] Ting M, Low JHM, Lee DPS, Fam J, Mahendran R, Kua EH, Kim JE. Impact of dietary counselling on cardiometabolic health, mental health and dietary quality in Singapore older women. Nutr Metab Cardiovasc Dis. 2025 Dec 24:104536. doi: 10.1016/j.numecd.2025.104536. Online ahead of print. PMID 41622098